CLINICAL TRIAL: NCT03136094
Title: Collaborative Hub to Reduce the Burden of Suicide Among Urban American Indian and Alaska Native Young Adults
Brief Title: Suicide in Urban Natives: Detection and Networks to Combat Events
Acronym: SUNDANCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Washington State University (Other); University of New Mexico (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 18-0186; U19MH113135 (NIH)
Record Dates: First submitted 2017-04-27; First posted 2017-05-02 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Suicide Prevention
Keywords: American Indian; Alaska Native; Youth and Young Adult; SBIRT
MeSH Terms: conditions — Suicide Prevention

STUDY DESIGN:
Intervention Model Description: The Investigators will conduct a randomized controlled trial to test the effectiveness of an augmented Screening, Brief Intervention, and Referral to Treatment (SBIRT) model that includes sending caring text messages for 12 months after an at-risk patient is identified.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will not be given details about how text messaging differs for the 2 study groups. Instead, patients will be told that the clinic is testing a program to support people who are having hard times, and that they will receive periodic text messages from the Site Coordinator for the next 12 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SBIRT+Usual Care (Placebo Comparator): The control arm of the trial will receive the usual care prescribed in the Screening, Brief Intervention and Referral to Treatment (SBIRT) model.
  Interventions: Behavioral: SBIRT+Usual Care
- SBIRT+12 (Experimental): The standard SBIRT model is augmented by a 12 month period following identification of suicide risk during which participants will receive caring text messages adapted from empirically-based, effective interventions for suicide prevention among American Indian and Alaska Native young adults.
  Interventions: Behavioral: SBIRT+12

INTERVENTIONS:
Behavioral: SBIRT+12 — The standard SBIRT model is augmented by a 12 month period following identification of suicide risk during which participants received caring text messages adapted from empirically-based, effective interventions for suicide prevention among American Indian and Alaska Native young adults.
  Arms: SBIRT+12
Behavioral: SBIRT+Usual Care — Patients receive usual SBIRT care
  Arms: SBIRT+Usual Care

SUMMARY:
This study compares the effectiveness of a program to detect and manage suicide risk among American-Indian and Alaska Native (AI/AN) youth. Half of the participants will receive caring text messages to reduce suicidal thoughts, attempts, and hospitalizations and to increase engagement, social connectedness, and resilience in at-risk youth. The other half will receive usual care that does not include the caring text messages.

DETAILED DESCRIPTION:
The study, "Suicide in Urban Natives: Detection and Networks to Combat Events," builds on Screening, Brief Intervention and Referral to treatment (SBIRT), carried out through the primary care setting, to detect and manage suicide risk. This approach is multilevel, targeting both the healthcare system and the individual, and links screening to existing mobile phone technologies shown to promote resilience and to tap the protective benefits of social connectedness. This Collaborative Hub will conduct a randomized control trial that compares the effectiveness of enhancing these SBIRT programs by sending caring text messages to reduce suicidal ideation, attempts, and hospitalizations, and to increase engagement, social connectedness, and resilience. The Investigators' long-term goal is to disseminate and translate the lessons learned into practical policy, organizational changes, and preventive innovations that optimize patient-centered health outcomes and ultimately reduce or eliminate the dramatic and tragic suicide-related health disparities among urban AI/AN youth and young adults.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as American Indian or Alaska Native;
* Screen positive for mild, moderate, or severe risk of suicidality (referred by a clinical provider);
* Have a text-enabled mobile phone;
* Willing to be contacted by text;
* Able to participate voluntarily;
* Speak and read English;
* Cognitively able to independently provide written informed consent

Exclusion Criteria:

* Under age 18
* In danger of imminent self-harm;
* Hospitalized

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 698 (Estimated)
Dates: Start 2020-03-15 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Suicidal Ideation | Baseline, 6 months, 12 months
  The 15-item Suicidal Ideation Questionnaire Jr. assesses frequency of suicidal thoughts in the past month. Item content ranges from general thoughts of death and wishes that one were dead to specific thoughts of self-injurious behavior. Responses are on a 7-point scale ranging from never to almost daily. Items are summed for a total score (range 0-90).
Change in Self-Reported Suicide Attempts | Baseline, 6 months, 12 months
  The investigators will use the interviewer-administered Suicide Attempt and Self-Injury Count to assess the method, intent, treatment received, and lethality for all suicide attempts over the respondent's lifetime.
Change in Hospitalizations and Behavioral Health Treatment | Baseline, 6 months, 12 months
  The investigators will assess self-reported hospitalizations over the previous 12 months with a measure of health service use previously applied to AI/ANs. It captures information on inpatient and outpatient medical care, emergency room visits, and use of traditional practices.

SECONDARY OUTCOMES:
Change in Social Connectedness | Baseline, 6 months, 12 months
  The investigators will assess social connectedness with the Interpersonal Needs Questionnaire, a validated measure of feelings of connectedness to others and of being a burden on others.
SBIRT Retention and Uptake of Referral to Therapy | 6 months, 12 months
  Retention will be measured as binary indicators of complete participation in the appropriate level of intervention determined during the initial in-person session with the behavioral therapist before enrollment in the study, and as uptake of therapy services for people who are referred to this level of care. For each participant, we will create a 3-category indicator of retention (full, partial, none).

CONTACTS AND LOCATIONS:
Overall Officials: Spero Manson, PhD, Principal Investigator — University of Colorado, Denver; Dedra Buchwald, MD, Principal Investigator — University of Washington
Locations (1):
- First Nations Community HealthSource, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herne MA, Bartholomew ML, Weahkee RL. Suicide mortality among American Indians and Alaska Natives, 1999-2009. Am J Public Health. 2014 Jun;104 Suppl 3(Suppl 3):S336-42. doi: 10.2105/AJPH.2014.301929. Epub 2014 Apr 22. PMID 24754665
- [Background] Mann JJ, Apter A, Bertolote J, Beautrais A, Currier D, Haas A, Hegerl U, Lonnqvist J, Malone K, Marusic A, Mehlum L, Patton G, Phillips M, Rutz W, Rihmer Z, Schmidtke A, Shaffer D, Silverman M, Takahashi Y, Varnik A, Wasserman D, Yip P, Hendin H. Suicide prevention strategies: a systematic review. JAMA. 2005 Oct 26;294(16):2064-74. doi: 10.1001/jama.294.16.2064. PMID 16249421
- [Background] Luoma JB, Martin CE, Pearson JL. Contact with mental health and primary care providers before suicide: a review of the evidence. Am J Psychiatry. 2002 Jun;159(6):909-16. doi: 10.1176/appi.ajp.159.6.909. PMID 12042175
- [Background] Beals J, Novins DK, Whitesell NR, Spicer P, Mitchell CM, Manson SM. Prevalence of mental disorders and utilization of mental health services in two American Indian reservation populations: mental health disparities in a national context. Am J Psychiatry. 2005 Sep;162(9):1723-32. doi: 10.1176/appi.ajp.162.9.1723. PMID 16135633
- [Derived] Morgan ER, Bogic M, Hebert L, Poole E, Tsosie N, Tsosie N, Garcia K, O'Leary M, Mettler R, Johnson G, Son-Stone L, Parker T, Buchwald D, Manson S. Caring Text Messages for Suicide Prevention in Urban American Indian Youth: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Sep 26;14:e71344. doi: 10.2196/71344. PMID 41004795